CLINICAL TRIAL: NCT00202163
Title: A Randomized Double-Blind Placebo-Controlled Study Comparing the Safety and Efficacy of Dehydroepiandrosterone (DHEA) or Testosterone Versus Placebo in Men With Sexual Dysfunction
Brief Title: ANDRO 2002: Dehydroepiandrosterone (DHEA) or Testosterone Versus Placebo in Men With Sexual Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Joe Downey, Centre Administrator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHEA-RCT
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Erectile Dysfunction
Keywords: ED; DHEA; testosterone
MeSH Terms: conditions — Erectile Dysfunction | interventions — Dehydroepiandrosterone; Testosterone

INTERVENTIONS:
Drug: DHEA
Drug: Testosterone

SUMMARY:
Androgen deficiency in the aging male is poorly understood. The objective of this study will be to determine the role of testosterone and DHEA in enhancing sexual interest and sexual performance.

DETAILED DESCRIPTION:
120 men with a diagnosis of Erectile dysfunction (ED) will be randomized to one of three arms in the study, DHEA (50 mg), testosterone [T] (80 mg) or placebo. Patients will be evaluated after starting blinded medication at 30 day intervals for a total of 90 days. Response will be evaluated with blood parameters, physical examination including rectal examination, validated questionnaires and global assessment scales.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction (ED)

Exclusion Criteria:

* Prior use of DHEA or T

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction

SECONDARY OUTCOMES:
Responder rates based upon questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Morales, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Advanced Urological Research, Kingston, Ontario, Canada